CLINICAL TRIAL: NCT06365723
Title: Effects of Walking in Greenspace and the Built Environment in Adults With Prediabetes: A Randomized Crossover Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: SPH-2023-32410
Record Dates: First submitted 2024-03-20; First posted 2024-04-15 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: PreDiabetes; Heart Rate Variability (HRV); Stress and Anxiety; Stress Biomarkers
Keywords: walking intervention; built environment; outdoor environment; prediabetes; stress; urban
MeSH Terms: conditions — Prediabetic State; Anxiety Disorders | interventions — Built Environment

STUDY DESIGN:
Intervention Model Description: The study is a randomized crossover trial with a 5-week washout period.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nature-based Walking then Built-environment/Commercial Walking (Experimental): People with prediabetes randomized to six weeks of nature-based walking followed by a five week washout, and then six weeks of built-environment/commercial-based walking
  Interventions: Behavioral: Nature-based Walking; Behavioral: Built-environment/Commercial Walking
- Built-environment/Commercial Walking then Nature-based Walking (Experimental): People with prediabetes randomized to six weeks of built-environment/commercial-based walking followed by a five week washout, and then six weeks of nature-based walking
  Interventions: Behavioral: Nature-based Walking; Behavioral: Built-environment/Commercial Walking

INTERVENTIONS:
Behavioral: Nature-based Walking — All participants will be asked to walk three to five times per week for 30-50 minutes per walk, totaling 150 min/week, at moderate intensity over a 6-week period in a designated nature-based, or 'green', urban environment.
Behavioral: Built-environment/Commercial Walking — All participants will be asked to walk three to five times per week for 30-50 minutes per walk, totaling 150 min/week, at moderate intensity over a 6-week period in a designated built-environment/commercial, or 'Gray', urban environment.

SUMMARY:
The goal of this randomized crossover trial is to compare the differences in psychological and physiological effects of walking in two different outdoor environments (urban/suburban commercial environments vs. urban/suburban nature areas/preserves) in adults with prediabetes. The main questions it aims to answer are:

* Do psychological measures of stress, anxiety, and affect improve more in one type of outdoor environment over the other?
* Do physiological measures of stress improve more in one type of outdoor environment over the other?

As this is a crossover trial, participants will serve as their own controls. Researchers will compare both the psychological and physiological effects walking in the two types of outdoor environments.

Participants will:

* Walk 150-minutes per week for six weeks in each of the two outdoor conditions.
* Visit the clinic four times, including before and after each six-week walking period.
* Collect saliva samples immediately proceeding or following the four clinic visits.
* Return to their pre-study level of physical activity for a 5-week washout period between each of the two walking interventions.

DETAILED DESCRIPTION:
Approximately 92 million U.S. adults (~38% of population) have prediabetes (PreD). Because people with PreD are at high risk CMD, they are a target population for diabetes prevention programs. The focus is people with PreD because of their high risk for developing CMD and large numbers, providing an opportunity to investigate behavioral and environmental approaches as preventive measures in a well-defined population. Urbanization affords challenges and opportunities to public health that include exposure to obesogenic environments, air pollution, and psychosocial stressors. In healthy adults suggest exposure to nature has health benefits relative to exposure to built environments. Hypothesized mechanisms for health benefits of Greenspace exposure include increased physical activity (PA), attention restoration, stress reduction, and reduced exposure to pollution. Many of the health benefits are associated with reduced psychological and physiological stress leading to better autonomic functioning as assessed by heart rate variability (HRV) and other biomarkers. Multiple studies suggest that PA and exposure to natural environments may act together to improve health. Yet, aside from our preliminary studies, we are not aware of any studies that examined how physical activity may interact with exposure to urban Greenspace ('Green') compared with built urban environments ('Gray'), to reduce stress and improve health. The purpose of this proposed study is to conduct a randomized crossover trial comparing differences in the psychosocial and physiological effects of walking in urban Green and Gray spaces in adults with PreD.

ELIGIBILITY:
Inclusion Criteria:

* 25-64 years old.
* Classified as overweight or obese with BMI 20.0-39.9 kg/m2 per self-report and a BMI of 20.0- 41.9 kg/m2 upon actual measure.
* Documentation* of a PreD diagnosis within one year of enrollment by physician or primary care provider based on lab tests showing a fasted blood glucose of 100-125 mg/dL, a 2-hour oral glucose tolerance test of 140-199 mg/dL, or an HbA1c level of 5.7%-6.49%271; OR a study screening lab value of HbA1C within the aforementioned range.
* Currently engaged in ≤100 min/week of moderate to vigorous exercise -confirmed via a 7-day activity recall.
* No exercise contraindications as assessed by the Physical Activity Readiness Questionnaire (PAR-Q) -this Questionnaire involves seven "yes" or "no" questions regarding an individual's health status. Answering "yes" to any one of these questions may require a prospective participant to acquire a written doctor's note stating they can safely participate in the trial's exercise intervention. The participant would not be enrolled until this doctor's note is received.
* Stable weight over the last 3 months (less than 10% change).
* Not currently pregnant, planning to become pregnant, or currently breastfeeding.
* Willing to maintain current dietary and exercise habits, aside from any changes to be made per the study exercise protocol.
* Must own a smartphone and be willing and able to download the Garmin Connect app
* Ability to speak and understand English.
* Any level of income
* Any race/ethnicity

Exclusion Criteria:

* Individuals <25 or >64: younger individuals may have not yet reached physiological maturity and in whom PreD prevalence is low; older individuals are more likely to have contraindications to PA and other comorbidities.
* BMI <20 or ≥42.
* Individuals with an HbA1c level <5.7% or >6.4%.
* Currently engaged in >100 min/wk of PA.
* Individuals with contraindications to exercise participation as indicated by the PAR-Q.
* A self-reported physical/mental disability that would prevent them from being able to adhere to the intervention.
* Past or current diagnosis of Diabetes (Type 1, 1.5 or 2) or use of diabetic medications (e.g. medications to control blood sugar)
* Any history of a cardiovascular disease event (e.g. heart attack, ablation, pacemaker, stroke)
* Current treatment for cancer or heart disease (lipid and hypertensive medications acceptable but will be tracked closely).
* Any change within the last 3 months, or anticipated changes, of any medications that would affect study outcomes (e.g. medications for lipids, blood pressure, anxiety, depression)
* The use of any medication that significantly interferes with the autonomic nervous system
* Current tobacco or nicotine users, or those who have quit within the last six months
* Excessive alcohol (on average>1 drinks/day for women and >2 drinks/day for men) or excessive recreational drug use (reported usage of once a week or more).
* Unstable weight over the last three months (>10% change).
* Those with major surgery planned or recent history of bariatric surgery (within last 2 years) or a history of other medical interventions that would interfere with study outcomes
* Currently within one-year postpartum, currently pregnant, or planning to become pregnant during the study period.
* Currently breastfeeding.
* Unwilling to comply with study randomization procedures.
* Unwilling to maintain current dietary and exercise habits, aside from any changes to be made per the study exercise protocol.
* Current participation in another interventional clinical trial.
* Previous randomization in this study.

Ages: 25 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 216 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Measure of Anxiety | Before and after each of the four assessment walks, which occur in weeks 4, 7, 15, and 18 (weeks 3 and 6 of each 6-week walking intervention).
  An Ecological Momentary Assessment of anxiety (rating level on a 0-10 point Likert scale) will be assessed pre/post each assessment walk.
Perceived stress assessment | Before and after each of the four assessment walks, which occur in weeks 4, 7, 15, and 18 (weeks 3 and 6 of each 6-week walking intervention).
  Perceived stress will be measured using an Ecological Momentary Assessment of stress (rating level on a 0-10 point Likert scale) will be assessed pre/post each assessment walk.
Mood assessment | Before and after each of the four assessment walks, which occur in weeks 4, 7, 15, and 18 (weeks 3 and 6 of each 6-week walking intervention).
  Mood will be evaluated using an Ecological Momentary Assessment of mood (i.e.. sadness, happiness, relaxation, mental energy, and physical energy) will be assessed pre/post each assessment walk (rating level on a 0-10 point Likert scale).
Restorativeness | Assessment given after each of the four assessment walks, which occur in weeks 4, 7, 15, and 18 (weeks 3 and 6 of each 6-week walking intervention).
  Assessing the restorativeness of the walked environment (using the perceived restorativeness scale) after each of the four assessment walks.

SECONDARY OUTCOMES:
Walking Heart Rate variability | Before, during, and after each of the four assessment walks, which occur in weeks 4, 7, 15, and 18 (weeks 3 and 6 of each 6-week walking intervention).
  Heart rate variability (HRV) will be measured before, during (within steady-state walking), and after each of the four assessment walks. We will use the Zephyr BioHarness and associated BioModule to complete these measurements. The a priori metric for analysis is the HRV during the walk between minutes 10 and 30.
Salivary cortisol levels | Within 7 days of each of the four clinic visits which occur before and after each of the 6-week walking interventions (i.e. study weeks 1, 7, 12 and 18).
  Saliva will be collected using the passive drool collection method at the following daily times: (1) immediately upon waking; (2) 30-45 minutes after waking; and (3) 14 hours after waking. Sampling times allow for calculation of the cortisol awakening response and diurnal decline in cortisol, metrics well correlated with health outcomes. Salivary cortisol will be assayed using validated ELISA assays
Ambient Particulate Matter | During each of the four assessment walks, which occur in weeks 4, 7, 15, and 18 (weeks 3 and 6 of each 6-week walking intervention).
  Ambient Particulate Matter will be assessed using the AirBeam3, a palm-sized air quality instrument that measures PM1, PM2.5, PM10, temperature, and relative humidity. It will be worn during each of the four assessment walks, measuring air-quality in real time as the participant is out on their walk.
CMD risk | At each of the four clinic visits which occur before and after each of the 6-week walking interventions (i.e. study weeks 1, 7, 12 and 18).
  CMD risk score will be computed as the average of the z-scores comprised of systolic blood pressure, and fasting blood glucose, insulin, triglycerides, and HDL-cholesterol (reverse scored).

OTHER OUTCOMES:
Resting Heart Rate Variability | At each of the four clinic visits which occur before and after each of the 6-week walking interventions (i.e. study weeks 1, 7, 12 and 18).
  Resting Heart rate variability (HRV) will be measured at the Baseline and Follow-up visits for each of the two study conditions (Weeks 1, 7, 12, and 18). We will use the Zephyr BioHarness and associated BioModule to complete these measurements.
Anxiety | At each of the four clinic visits which occur before and after each of the 6-week walking interventions (i.e. study weeks 1, 7, 12 and 18).
  Anxiety will be assessed at each of the four clinical visits (occurring before and after each of the 6-week walking interventions) using the PROMIS Anxiety 8a.
CMD-Risk Mediation | Throughout the study, up to 18 weeks.
  The extent to which physiological, psychological, and air pollution measures mediate the differential impact of Green versus Grey walking on CMD-risk using regression-based mediation models.
Stress | At each of the four clinic visits which occur before and after each of the 6-week walking interventions (i.e. study weeks 1, 7, 12 and 18).
  Stress will be assessed at each of the four clinical visits (occurring before and after each of the 6-week walking interventions) using the Perceived Stress Scale.
Affect | At each of the four clinic visits which occur before and after each of the 6-week walking interventions (i.e. study weeks 1, 7, 12 and 18).
  Affect will be assessed at each of the four clinical visits (occurring before and after each of the 6-week walking interventions) using the PROMIS Affect 15a.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Pereira, PhD, Principal Investigator — University of Minnesota
Locations (3):
- United States (3):
  - Lake Forest Hospital, Lake Forest, Illinois
  - Central DuPage Hospital, Winfield, Illinois
  - Epidemiological Clinical Research Center, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study website for more information and contacts. — https://www.sph.umn.edu/research/projects/wonder-study/